CLINICAL TRIAL: NCT05261217
Title: Three-Dimensional Evaluation of the Airway Space After Distalization in Adults Using Carrière Motion Appliance: Cone Beam Computed Tomographic Study
Brief Title: Three-Dimensional Evaluation of the Airway Space After Distalization in Adults Using Carrière Motion Appliance
Acronym: CBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Heba Allah Ahmed Ahmed ELghawy, Heba Allah Ahmed Ahmed Elgahawy, Suez Canal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192/2019
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Orthodontic Appliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The motion 3D II appliance (Experimental): using The motion 3D II appliance on treating Class II orthodontic
  Interventions: Device: The motion 3D II appliance

INTERVENTIONS:
Device: The motion 3D II appliance — The motion 3D II appliance treating class II malocclusion

SUMMARY:
Class II malocclusion is quite possibly most continuous treatment issues confronting orthodontists, addressing just about 33% malocclusions. connection between II malocclusion decreased pharyngeal aviation route measurements has been accounted for in writing. few treatment alternatives have been endeavored address this malocclusion, one those choices is distalize maxillary back without extraction treatment. In 2004 another machine presented Luis Carrière conveying his name, called Carrière Motion apparatus. Nonetheless, so far RCT in orthodontic writing assessed impact this machine elements aviation route.

The point this examination assess impact this machine upper aviation route CBCT pictures in treatment post-pubertal patiets dental II malocclusion. near report led comprising 18 members age range from 18-30 years age. treatment impacts assessed radiographically utilizing pre post-distalization CBCT pictures after I connection has been reached. three dimentional investigation performed contemplate impacts distalization upper aviation route. gathered information then genuinely broke down for treatment changes among pre post-distalization.

DETAILED DESCRIPTION:
Patients selected from outpatient center at Department Orthodontics, Faculty Oral Dental Medicine, Suez Canal University. Research Ethical Committee Faculty Oral Dental Medicine, Suez Canal University endorsed this investigation. Patients educated about methodology shown logical, enlivened recordings.

3. Incorporation standards:

The chose patients had met accompanying models:

a) Adults full lasting dentition matured from (18-30). b) Dental II malocclusion beginning from half unit three quarter unit II relationship reciprocally where treatment plan did exclude extraction in upper curve.

c) A ordinary skeletal maxilla typical or gentle direct retrognathic mandible. d) Normal or flat development design. e) All patients ought have great oral cleanliness ought consent inspiration directions give sensible forecast.

f) Absence ejected maxillary third molars. g) The patients should be liberated from any foundational illness or medical conditions.

4. Prohibition models:

1. Patients set experiences any genuine injury or medical procedure orofacial district.
2. sex inclination.
3. No history orthodontic treatment subjects.
4. No history obstructive breathing issues. 5-Methodology: 5.1 Preoperative intercession:

A Medical History Questionnaire:

A clinical filled patients bar any patients who might be experience ill effects any fundamental illness. Besides, patients checked ear nose throat expert affirm shortfall any aviation route problem.

5.2 Dental Case History Clinical Examination: A total dental case history acquired from every quiet patients analyzed clinically submitted both extraoral intraoral assessment. patients checked meet incorporation measures recently referenced. chose patients who met rules, alluded Periodontal Department centers for additional improvement oral cleanliness Restorative Department Clinics for any necessary fillings lastly alluded Oral Maxillofacial Surgery Department for extraction third maxillary molars in case they completely ejected in oral cavity.

5.3 Patients' Records: The accompanying records acquired from every understanding before endless supply treatment time, 5.3.1 Photographs For every tolerant bunch 4 extraoral 5 intraoral photos taken 5.3.2 Orthodontic Study Models All patients submitted upper lower impressions utilizing alginate impressionA material. wax wafer chomp additionally acquired. Impressions poured promptly utilizing extra hard stone model bases appropriately framed managed orthodontic norms 5.3.3 Cone Beam Computed Tomography: The chose patients submitted two CBCT examines; one pre-usable another after finish distalization utilizing Carrière Motion machine. CBCT pictures procured utilizing SOREDEX SCANORA 3D present in radiology office in Faculty Dentistry Suez Canal University. CBCT examining is performed producer's convention similar administrator. boundaries CBCT set suggestion assembling

ELIGIBILITY:
Inclusion Criteria:

Dental II malocclusion beginning from half unit three quarter unit II relationship reciprocally where treatment plan did exclude extraction in upper curve.

A ordinary skeletal maxilla typical or gentle direct retrognathic mandible. Normal or flat development design. All patients ought have great oral cleanliness ought consent inspiration directions give sensible forecast.

Absence ejected maxillary third molars. The patients should be liberated from any foundational illness or medical conditions.

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Cone Beam Computed Tomography | nine months
  CBCT with Nasopharyngeal Airway Nasopharyngeal Airway Volume Oropharyngeal Airway
  Oropharyngeal Airway volume Hypopharyngeal Airway Hypopharyngeal Airway volume parameters

CONTACTS AND LOCATIONS:
Overall Officials: Heba Allah ELghawy, Bachlor, Principal Investigator — Suez Canal University
Locations (1):
- Faculty of dentistry, Suez canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No